CLINICAL TRIAL: NCT02671019
Title: Comparing Effectiveness and Costs of Internet-based Treatment for Problematic Alcohol Use and Face-to-face Treatment in Addiction Care: A Randomized Controlled Trial
Brief Title: Effectiveness and Costs of Internet-based Treatment for Harmful Alcohol Use and Face-to-face Treatment in Addiction Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Kristina Sinadinovic, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1758-31/2
Record Dates: First submitted 2016-01-11; First posted 2016-02-02 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Use Disorders
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based treatment (Experimental): A five-module Internet-based treatment program for harmful alcohol use (including therapist support) based on Motivational Interviewing, Cognitive Behavioral Treatment and Relapse prevention, focusing on: Motivation to change harmful alcohol use, defining a goal for the treatment, self-control strategies, risk situations, planning alternative behaviors and relapse prevention.
  Interventions: Behavioral: Guide to better alcohol habits
- Face-to-face treatment (Active Comparator): Same treatment content as in the Internet-based treatment delivered via face-to-face treatment sessions in specialized addiction treatment.
  Interventions: Behavioral: Guide to better alcohol habits

INTERVENTIONS:
Behavioral: Guide to better alcohol habits — A treatment for harmful alcohol use based on Motivational Interviewing, Cognitive Behavioral Treatment and Relapse prevention, focusing on: Motivation to change harmful alcohol use, defining a goal for the treatment, self-control strategies, risk situations, planning alternative behaviors and relapse prevention.

SUMMARY:
The purpose of this trial is to compare the effectiveness and costs of a five-module Internet-based treatment program (including therapist support) for harmful alcohol use with the effectiveness and cost of the same treatment content delivered face-to-face in specialized addiction treatment. The hypotheses to be tested through this trial are that:

1. The Internet-based treatment program (including therapist support) is as effective (reducing alcohol consumption) as the same treatment content delivered face-to-face in specialized addiction treatment.
2. The Internet-based treatment program (including therapist support) is associated with lower cost per treated individual in relation to the achieved effects (in terms of reduced alcohol consumption) compared with the same treatment content delivered face-to-face in specialized addiction treatment.

The design is a two-armed randomized controlled trial, and outcomes are measured in terms of changes in alcohol consumption, problematic alcohol use as well as alcohol dependence, depression, anxiety, quality of life and costs for the treatments. A minimum of 350 participants will be recruited and randomized into two groups:

Intervention group 1: All participants in this group will have access to the five-module Internet-based treatment program for harmful alcohol use and have access to a therapist with training in psychotherapy (CBT) who assists and counsels the participant throughout the program.

Intervention group 2: All participants in this group will attend five face-to-face treatment sessions in specialized addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* 16 points on Alcohol Use Disorders Identification Test or at least 3 criteria on the International Classification of Diseases (ICD-10) for Alcohol Dependence
* Resident in Stockholm County

Exclusion Criteria:

* Lack of understanding of the Swedish language.
* Doctor's assessment that there is a risk for severe withdrawal symptoms, risk for suicide or mental illness requiring separate care.
* Doctor's assessment that there is a need for medication for alcohol dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of standard alcohol units consumed in the past 7 days measured with Time Line Follow Back method | 3 months post-randomization

SECONDARY OUTCOMES:
Number of standard alcohol units consumed in the past 7 days measured with Time Line Follow Back method | 6 months post-randomization
Number of standard alcohol units consumed in the past 7 days measured with Time Line Follow Back method | 12 months post-randomization
Number of standard alcohol units consumed in the past 7 days measured with Time Line Follow Back method | 24 months post-randomization
Alcohol Use Disorders Identification Test score | 3 months post-randomization
Alcohol Use Disorders Identification Test score | 6 months post-randomization
Alcohol Use Disorders Identification Test score | 12 months post-randomization
Alcohol Use Disorders Identification Test score | 24 months post-randomization
Number of criteria for alcohol dependence according to International Classification of Diseases - 10 | 3 months post-randomization
Number of criteria for alcohol dependence according to International Classification of Diseases - 10 | 6 months post-randomization
Number of criteria for alcohol dependence according to International Classification of Diseases - 10 | 12 months post-randomization
Number of criteria for alcohol dependence according to International Classification of Diseases - 10 | 24 months post-randomization
Number of criteria for alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - V | 3 months post-randomization
Number of criteria for alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - V | 6 months post-randomization
Number of criteria for alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - V | 12 months post-randomization
Number of criteria for alcohol dependence according to Diagnostic and Statistical Manual of Mental Disorders - V | 24 months post-randomization
Number of days absent from work due to illness | 3 months post-randomization
Number of days absent from work due to illness | 6 months post-randomization
Number of days absent from work due to illness | 12 months post-randomization
Number of days absent from work due to illness | 24 months post-randomization
Score on Montgomery-Åsberg Depression Rating Scale | 3 months post-randomization
Score on Montgomery-Åsberg Depression Rating Scale | 6 months post-randomization
Score on Montgomery-Åsberg Depression Rating Scale | 12 months post-randomization
Score on Montgomery-Åsberg Depression Rating Scale | 24 months post-randomization
Score on Generalised Anxiety Disorder 7-item scale | 3 months post-randomization
Score on Generalised Anxiety Disorder 7-item scale | 6 months post-randomization
Score on Generalised Anxiety Disorder 7-item scale | 12 months post-randomization
Score on Generalised Anxiety Disorder 7-item scale | 24 months post-randomization
Score on EQ-5D measuring the quality of life | 3 months post-randomization
Score on EQ-5D measuring the quality of life | 6 months post-randomization
Score on EQ-5D measuring the quality of life | 12 months post-randomization
Score on EQ-5D measuring the quality of life | 24 months post-randomization
Cost for treatment | 3 months post-randomization
Cost for treatment | 6 months post-randomization
Cost for treatment | 12 months post-randomization
Cost for treatment | 24 months post-randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden